CLINICAL TRIAL: NCT02454036
Title: Psychological Changes in Cancer Patients Receiving a Biobehavioral Intervention: A Program Evaluation
Brief Title: Biobehavioral Intervention in Gynecologic Oncology Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rachel Miller (Other)
Responsible Party: Sponsor-Investigator, Rachel Miller, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-GYN-02-MCC; R25CA163197 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vulva
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BBI Intervention (Experimental): Biobehavioral Intervention
  Interventions: Behavioral: BBI intervention

INTERVENTIONS:
Behavioral: BBI intervention — Psychological intervention designed to reduce stress and enhance quality of life
  Other Names: Biobehavioral Intervention

SUMMARY:
Baseline self-report outcome measures will be completed and additional assessments will occur mid-treatment , post-treatment , 3 months following completion of all sessions, and 6 months following completion of all sessions. Patients and therapists will complete the evaluation measures in private (at home, in an office).

At the University of Kentucky Markey Cancer Center, BBI treatment is offered in group and individual formats. The course of individual treatment varies and group treatment consists of 10 1.5-hour weekly sessions in the "intensive" phase, followed by 2 1.5-hour bi-weekly maintenance sessions. Individual treatment is one-on-one. In group treatment, there are typically 6-12 patients per group and 1 or 2 therapists. The intervention helps patients to learn adaptive coping strategies and how to apply them to daily stressors. Additional content discusses use of seeking information, enhancing social support, enhancing body esteem and intimacy, and maintaining positive changes.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Stage I-IV gynecologic cancer (including ovarian, uterine, cervical, vulvar, or vaginal cancer)
* Undergoing active treatment or in remission and undergoing active surveillance; age ≥21 and ≤80
* Able to speak/read English.

Exclusion Criteria:

* Concurrent diagnosis of organic brain syndrome, dementia, mental retardation
* Non-English speaking, or significant sensory deficit
* Major mental illness (e.g., schizophrenia, psychotic disorder).

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Emotional distress as measured by Profile of Mood States score | Up to 6 months following completion of treatment
Cancer specific traumatic stress as measured the by Impact of Events Scale score | Up to 6 months following completion of treatment
Social support as measured by the Perceived Social Support from Family score | Up to 6 months following completion of treatment
Physical activity as measured by the Godin-Shepard Leisure-Time Physical Activity Questionnaire score | Up to 6 months following completion of treatment
Dietary habits as measured by the Food Habits Questionnaire | Up to 6 months following completion of treatment
Sexual functioning as measured by the Sexual Experience Scale score | Up to 6 months following completion of treatment
Pain as measured by the Brief Pain Questionnaire score | Up to 6 months following completion of treatment
Fatigue as measured by the Fatigue Severity Index score | Up to 6 months following completion of treatment
Sleep as measured by the Pittsburg Sleep Quality Index | Up to 6 months following completion of treatment

SECONDARY OUTCOMES:
Patient-reported evaluation of the BBI as measured by the Evaluation of Topics score | Up to 6 months following completion of treatment
Therapist-reported fidelity/Usage of BBI as measured through logs | Up to 6 months following completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Miller, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States